CLINICAL TRIAL: NCT00158145
Title: Longitudinal Study of Prostate, Lung, Colon, and Ovarian Cancer (PLCO) Screen Trial
Brief Title: Assessing the Variability Over Time of Tobacco Carcinogen Biomarkers in Smokers - 2
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Tim Church, University of Minnesota
Other Study IDs: NIDA-13333-2; P50-13333-2; DPMC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-06

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood samples.

SUMMARY:
Lung cancer is the leading cause of cancer death in the United States. Currently it remains impossible to predict which smokers will get cancer. Each puff of a cigarette delivers a mixture of over 60 known carcinogens. Biomarkers that quantify carcinogen levels and metabolism are a useful tool and available to use. The purpose of this study is to assess the variability of tobacco smoke carcinogen biomarker levels over one year in a group of smokers.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the United States. Approximately 90% of lung cancer is caused by cigarette smoking. While most lung cancer cases occur in smokers or ex-smokers, only 15-25% of smokers will get lung cancer. Currently it remains impossible to predict which smokers will get cancer.

Each puff of a cigarette delivers, along with nicotine, a mixture of over 60 known carcinogens. Most of these carcinogens require metabolic activation before they can negatively affect cell DNA and cause cancer. Biomarkers that quantify carcinogen levels and metabolic activity of carcinogens are a useful tool and available to use. The purpose of this study is to assess the variability of tobacco smoke carcinogen biomarker levels over one year in a group of smokers.

This longitudinal observational study will involve a repeated measure analysis of 6 different tobacco carcinogen biomarkers. Fifty current smokers who intend to continue smoking for the duration of the study will be recruited through advertisements. Participants will be compensated for their time. Blood samples will be collected every two months for one year. All samples will be analyzed for the 6 different carcinogen biomarkers and individual variability in biomarker levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Currently smokes
* Intends to continue smoking for the 12 months following enrollment

Exclusion Criteria:

* Unstable physical or mental condition

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cigarette smokers
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States